CLINICAL TRIAL: NCT01433939
Title: Position Changes During Colonoscope Insertion Increases Patient Comfort: a Prospective Trial
Brief Title: Position Changes During Colonoscope Insertion Increases Patient Comfort
Status: Completed | Type: Observational
Sponsor: Jennifer Telford (Other)
Responsible Party: Sponsor-Investigator, Jennifer Telford, Clinical Assistant Professor, University of British Columbia
Organization: University of British Columbia (Other)
Other Study IDs: H11-01597
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Colonoscopy Technique
Keywords: colonoscopy; position changes; patient comfort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators wish to study the effects of position changes during colonoscope insertion on patient comfort. The investigators hypothesize that early position changes would reduce colonoscope loop formation and patient discomfort.

ELIGIBILITY:
Inclusion Criteria:

* age 19 years or older
* outpatient colonoscopy

Exclusion Criteria:

* inpatient
* unable to provide informed consent
* previous bowel resection, inflammatory bowel disease
* musculoskeletal disorder or other mobility issues limiting effective patient position changes.
* inadequate bowel preparation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to gastroenterologists for colonoscopy.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05-25 (Actual); Study Completion 2015-05-25 (Actual)

PRIMARY OUTCOMES:
Intensity and frequency of abdominal pain | 30min
  Abdominal pain during colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Telford, MD, Principal Investigator — The University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada